CLINICAL TRIAL: NCT00367341
Title: Imaging Predictors of Treatment Response in Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Helen Mayberg, Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00026176
Record Dates: First submitted 2006-08-18; First posted 2006-08-22 (Estimated); Results first posted 2014-01-09 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder
Keywords: Depression, Treatment, Imaging
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Cognitive Behavioral Therapy; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Escitalopram (Other)
  Interventions: Drug: escitalopram
- Cognitive Behavioral Therapy (Other)
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: escitalopram — Participants will receive treatment with escitalopram for 12 weeks.
  Other Names: Lexapro
  Arms: Escitalopram
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT will include 16 1 hour sessions provided over 12 weeks.
  Other Names: Talk Therapy
  Arms: Cognitive Behavioral Therapy

SUMMARY:
While there are many effective options for treating a major depressive episode, there are no clinical markers that predict the likelihood of remission with an initial trial of either an antidepressant medication or psychotherapy. More critically, there are also no reliable predictors that might anticipate failure to such standard treatments either alone or in combination. This project will characterize imaging-based brain subtypes that distinguish groups of depressed patients who later remit or not to SSRI pharmacotherapy or cognitive behavior therapy (CBT), respectively. To define these subtypes, a prospectively-treated cohort of 100 patients will be randomized to receive either escitalopram (s-CIT) or CBT for the first 12 weeks, with non-remitters to either first treatment crossed over to receive an additional 12 weeks of treatment with combined treatment. Non-remitters to both treatments will thus define a relatively treatment resistant third subgroup. Resting-state 18F-fluoro-deoxyglucose (FDG) positron emission tomography (PET) scans will be acquired prior to initiating antidepressant therapy, with pre-treatment scan patterns associated with three possible outcomes (CBT remission, s-CIT remission, and non-remission to both) assessed using multivariate analytic methods. A second PET scan, acquired early in the treatment course, will be used to assess the likelihood of response to the specific treatment first assigned. The proposed studies are a first step towards defining brain-based biomarkers predictive of differential treatment outcome in major depression; most critically, patterns distinguishing patients at risk for treatment resistance. Identification of such biomarkers has additional implications for future testing of novel therapies in patients with distinct brain signatures, including development of evidence-based treatment algorithms for individual patients.

DETAILED DESCRIPTION:
SPECIFIC AIMS Aim 1. To define baseline regional glucose metabolic patterns (measured using FDG PET) associated with differential clinical remission to each of two well-established, randomly delivered first-line antidepressant treatments-the SSRI escitalopram (s-CIT) or cognitive behavioral therapy (CBT) with cross-over treatment for non-remitters (sequential course of treatment model).

Aim 2. To define metabolic change patterns, occurring early in the course of both s-CIT and CBT, associated with successful and unsuccessful clinical remission to each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 60. (no subjects with first episode over age 50. This is an attempt to exclude patients with 'vascular depression' who have a potentially different pathophysiology and treatment response compared to idiopathic MDD.
* DSM-IV criteria for unipolar Major Depressive Disorder.
* HAM-D (24 item) score >/= 18 at Screening, >/= 15 at Baseline.
* Co-morbid conditions (other than those listed under exclusion criteria below) will be accepted as long as MDD is the primary diagnosis (based on predominance and sequential development of symptoms).
* Acceptable method of birth control (oral contraceptives, Depo-Provera, Norplant, condoms with spermicide. A vasectomy is acceptable in the framework of a stable monogamous relationship. Sexually inactive women must agree to contraception if they become sexually active during the study.
* Educational level, degree of understanding and reliability so that participation is feasible.
* Informed consent to participate and comply in the study.

Exclusion Criteria:

* Known neurological disorders or documented head injury.
* Serious and unstable medical illnesses including diabetes, cardiovascular disease and cancer.
* Medical conditions with known mood changes (endocrine, autoimmune disorders)
* Co-morbid DSM-IV Axis I Diagnoses

  1. Lifetime history of Bipolar Disorder, Schizophrenia, and other Psychotic Disorders, or Obsessive Compulsive Disorder
  2. Alcohol abuse or dependence within the past six months, psychoactive substance abuse or dependence within the past six months.
  3. Clinical evidence of a severe Personality Disorder that would impede participation or completion of a controlled trial.
* ECT within the past 6 months.
* Previous failure to achieve a much improved status on CGI-Improvement (the equivalent of >50% symptom reduction) with a course of CBT (defined as a minimum of 8 sessions during 8 weeks of a specified manual-driven therapy by a CBT trained therapist) or escitalopram (defined as a minimum of 6 weeks with the dose of 10 mgs achieved for at least 2 weeks)
* Use of concomitant medications with the exception of:

  1. Maintenance/prophylactic meds for stable medical conditions
  2. Ambien 5-10 mgs may be prescribed for occasional use (up to a single dose a week for insomnia, as long as it is not the night before a clinic visit, PET/fMRI study or ratings.
  3. Antidepressants will be discontinued for 7 days prior to the screening visit, which will be a minimum of a week before the baseline scan (5 weeks for fluoxetine, protryptyline).
* Current treatment with weekly individual or group psychotherapy targeted at the depressive symptoms, including psychodynamic, interpersonal or cognitive-behavioral.
* Currently responding to medication treatment, without clinical reasons to change (e.g. side effects). Will not enroll a subject who wishes to discontinue an effective treatment for the sake of participation in the research.
* Woman who are pregnant, breast feeding or intending to become pregnant during the course of the study.
* Contraindications for MRI: pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2006-08; Primary Completion 2011-08 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Mayberg, M.D., Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Result] McGrath CL, Kelley ME, Holtzheimer PE, Dunlop BW, Craighead WE, Franco AR, Craddock RC, Mayberg HS. Toward a neuroimaging treatment selection biomarker for major depressive disorder. JAMA Psychiatry. 2013 Aug;70(8):821-9. doi: 10.1001/jamapsychiatry.2013.143. PMID 23760393
- [Derived] McGrath CL, Kelley ME, Dunlop BW, Holtzheimer PE 3rd, Craighead WE, Mayberg HS. Pretreatment brain states identify likely nonresponse to standard treatments for depression. Biol Psychiatry. 2014 Oct 1;76(7):527-35. doi: 10.1016/j.biopsych.2013.12.005. Epub 2013 Dec 19. PMID 24462230
- See also: website with study information — http://www.emoryclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram: escitalopram : Participants will receive treatment with escitalopram for 12 weeks.
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) : CBT will include 16 1 hour sessions provided over 12 weeks.
Period: Overall Study
Arm/Group | Escitalopram | Cognitive Behavioral Therapy
Started | 42 | 40
Completed | 40 | 40
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 40 | 82
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (6.8) | 42.2 (9.5) | 41.68 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 16 | 18 | 34
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82

OUTCOME MEASURES:

1. Primary Outcome: Remission Defined as Hamilton Depression Rating Scale-17 Score of Less Than or Equal to 7 at 12 Weeks
Description: # of study participants with Hamilton Depression-17-item score less than or equal to 7.
Time Frame: Measured at week 12
Population: completed study participants in 12-week-trial
Measure: Number; unit: participants
Arm/Group | Escitalopram | Cognitive Behavioral Therapy
Number analyzed (Participants) | 32 | 31
participants | 12 | 12

2. Secondary Outcome: Response Defined as 50% Change in Hamilton Depression Rating Scale-17 Score at 12 Weeks
Description: Number of participants with a 50% change from Baseline on the Hamilton Depression Rating Scale-17-item score
Time Frame: Measured at week 12.
Population: completers
Measure: Number; unit: participants
Arm/Group | Escitalopram | Cognitive Behavioral Therapy
Number analyzed (Participants) | 32 | 31
participants | 18 | 18

ADVERSE EVENTS:
Arm/Group | Escitalopram | Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 33/42 | 21/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=42) | Cognitive Behavioral Therapy (N=40)
diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2)
fatigue (General disorders) | 5 (5) | 2 (2)
flu (Infections and infestations) | 3 (3) | 0 (0)
dizziness (General disorders) | 5 (5) | 0 (0)
dry mouth (General disorders) | 3 (3) | 0 (0)
headache (General disorders) | 14 (14) | 4 (4)
indigestion (Gastrointestinal disorders) | 4 (4) | 2 (2)
nausea (General disorders) | 10 (10) | 4 (4)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
stomach cramps (Gastrointestinal disorders) | 0 (0) | 2 (2)
constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)
insomnia (General disorders) | 7 (7) | 0 (0)
decreased libido (General disorders) | 6 (6) | 0 (0)
sedation (General disorders) | 11 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No